CLINICAL TRIAL: NCT03749044
Title: Aspirin Patterns of Use and Adherence for Prevention of Preeclampsia in SLE Pregnancies
Brief Title: ASA Patterns for Prevention of Preeclampsia in SLE Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of Calgary (Other); University of Toronto (Other); Dalhousie University (Other); University of British Columbia (Other); University of Manitoba (Other); University Health Network, Toronto (Other); Laval University (Other)
Responsible Party: Principal Investigator, Evelyne Vinet, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASA Pattern MP-37-2018-3915
Record Dates: First submitted 2018-10-23; First posted 2018-11-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia; Pregnancy Complications; Systemic Lupus
Keywords: Adverse Pregnancy Outcomes; SLE; Aspirin Adherence
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Educational Tool (Experimental): At the baseline visit, after having responded to the questionnaire, participants in the education arm will be given the patient educational tool.
  Interventions: Other: Patient Educational Tool
- Standard of Care (No Intervention): Subjects in the standard of care arm will not receive the patient educational tool. If participants ask specific questions on pregnancy complications and/or preeclampsia, the clinicians will provide relevant information as they judge appropriate, but without handing out the patient educational tool.

INTERVENTIONS:
Other: Patient Educational Tool — This tool is a modified version of the patient educational sheet elaborated and validated by You et al in collaboration with the Preeclampsia Foundation. This patient educational sheet graphically defines preeclampsia and its. A licensing agreement has been obtained from the Preeclampsia Foundation, with the rights to modify the educational tool for this RCT. The SLE-specific educational tool will consist in a sheet displaying the previously developed patient educational form on the recto. However, on the verso of the sheet, SLE-specific information related to the risk of preeclampsia in SLE pregnancies and the estimated efficacy of ASA in reducing preeclampsia risk in women at high risk are displayed.
  Arms: Patient Educational Tool

SUMMARY:
Preeclampsia is a serious maternal condition affecting up to 5% of pregnancies from the general population and up to 30% of lupus pregnancies. Aspirin (acetylsalicylic acid- ASA) has been shown to reduce the risk of preeclampsia, by half, in women at high risk. Therefore, it is recommended that health professionals initiate aspirin early during pregnancy in women with lupus. Despite this recommendation, there are currently no studies of aspirin in women with lupus for this indication. This is a critical knowledge gap as aspirin could potentially have a large benefit in this high-risk population.

The investigator will perform a RCT to evaluate the effect of a specifically designed patient educational tool on preeclampsia knowledge and ASA adherence in pregnant women with SLE.

The research efforts will improve reproductive health of SLE women and the outcomes of offsprings.

DETAILED DESCRIPTION:
The goal is to help improve counselling and ASA adherence for preeclampsia prevention in pregnant women with SLE. This study could offer the ideal setting for the conduct of a future study assessing the efficacy of ASA for prevention of placenta-mediated complications in SLE pregnancies.

For this trial, the investigator will recruit pregnant women with a SLE diagnosis based on the SLICC classification criteria, followed at the 6 Canadian SLICC centres (located in Toronto, Montreal, Halifax, Quebec, Winnipeg, and Calgary), at TRIO Fertility in Toronto and at Mary Pack Arthritis Centre, in Vancouver. Consecutive pregnant women speaking English or French and providing informed consent and meeting eligibility criteria will be recruited until the 12th gestational week. Investigator will only include one pregnancy per study subject in the study analyses. Investigator will include all single intrauterine pregnancies, occurring in women between the ages of 18-45 years, regardless of disease manifestations, level of disease activity, and medication exposures. Of note, all Canadian subjects recruited in the LEGACY cohort will be eligible to participate in this study.

Study subjects will be randomized in a 1:1 ratio to either the patient educational tool or standard of care. Individual subject randomization will be performed through a central web-based randomization system, using stratified blocked randomization with randomly selected block sizes.

For all study subjects, data will be obtained at baseline on demographics (maternal age, ethnicity, education, occupation), co-morbidities (e.g. hypertension, diabetes, chronic kidney disease, etc), alcohol and tobacco use, SLICC classification criteria, SLICC/ACR damage index (SDI), detailed lupus nephritis history (date of onset, lupus nephritis class as per biopsy if available, date of last renal flare), prior placenta-mediated complications (i.e. gestational hypertension, preeclampsia, eclampsia, small for gestational age neonate, stillbirth) and past/current medications.

Information on ASA including date of initiation, dosage, over-the-counter use, indication, and adherence will be recorded. Investigator will measure ASA adherence using the "Adherence to Refills and Medications Scale (ARMS)", which is a validated self-reported questionnaire developed for patients with chronic diseases with low literacy. It includes 12 short and simple questions, each scored 1 ("always") to 4 ("never"), and the total ranges from 12 to 48, with lower scores indicating higher levels of reported adherence. The investigator will define adherence as a continuous variable using the ARMS score, which has been shown to strongly correlate with both pill counts, pharmacy refills, and therapy response. Investigator will also record ASA adherence using a visual analogue scale.

Investigator will measure disease activity using the SLEPDAI. Investigator will also obtain data on BP, weight and height, renal function, urine microscopy, and UPCR. Autoantibodies, such as aPL antibodies, will be assessed locally at each centre and reported according to the centre specific normal ranges.

A 20-item questionnaire will be administered evaluating patient knowledge related to preeclampsia including both closed- and open-ended questions regarding the implications of preeclampsia, the symptoms associated with the syndrome, the role of ASA for its prevention, and the proper actions that should be taken if a patient experiences preeclampsia symptoms. The questionnaire will be scored by 2 independent investigators, calculating the percentage of correct responses. Once the questionnaire is completed at the baseline visit, results or correct answers will not be communicated to participants.

At the baseline visit, after having responded to the questionnaire, participants in the education arm will be given the patient educational tool. This tool is a modified version of the patient educational sheet elaborated and validated by You et al. in collaboration with the Preeclampsia Foundation. This patient educational sheet graphically defines preeclampsia and its complications and has been shown to substantially improve patient knowledge related to preeclampsia in a prior RCT, as mentioned previously. A licensing agreement from the Preeclampsia Foundation has been obtained, with the rights to modify the educational tool for this RCT. The SLE-specific educational tool will consist in a sheet displaying the previously developed patient educational form on the recto. However, on the verso of the sheet, SLE-specific information related to the risk of preeclampsia in SLE pregnancies and the estimated efficacy of ASA in reducing preeclampsia risk in women at high risk are displayed. The graphical display of the SLE-specific content has been optimized in consultation with relevant end-users.

Subjects in the standard of care arm will not receive the patient educational tool. If participants ask specific questions on pregnancy complications and/or preeclampsia, the clinicians will provide relevant information as judged appropriate, but without handing the patient educational tool.

At each study centre, investigators will complete a survey on the current practice of both rheumatologists and obstetricians regarding preeclampsia education and counselling of their SLE patients to gain insights into the standard of care at each site. The survey will be updated every 6 months. Of note, none of the sites have for standard of care of administering the Preeclampsia Foundation educational tool.

Patients will be reassessed in the 2nd (between 20-24 weeks), 3rd (between 30-34 weeks) trimesters, and in postpartum. At these visits, the investigator will record current medication use, including ASA initiation, dosage, indication for use, and adherence using the ARMS. In addition, the investigator will update information on placenta-mediated complications, disease manifestations, disease activity, BP, serum creatinine, urine microscopy and UPCR. The investigator will reassess patient preeclampsia knowledge at subsequent visits in both study groups by administering the same preeclampsia knowledge questionnaire to determine whether any enhancement of knowledge is retained. Informed consent has been obtain to include data collected from this RCT in the LEGACY biobank.

Statistical Analyses Patterns of ASA Use in SLE Women Receiving Standard of Care: Descriptive statistics will be used to measure the prevalence of ASA use at baseline and compare the prevalence of use across all trimesters in subjects receiving standard of care. In addition, the investigator will determine the proportion of patients who initiated ASA during pregnancy as well as the proportion of subjects already on ASA prior to pregnancy, exploring indications of use. The investigator will also measure the frequencies of dosage used (i.e. 80 mg, 160 mg, and 325 mg). Exploratory analyses will examine correlates of ASA initiation, as well as ASA non-adherence, during pregnancy in both groups using a bivariate regression analysis estimated with the generalized estimating equation method, evaluating the following baseline covariates while adjusting for educational tool exposure: maternal age, race/ethnicity, obesity, aPL autoantibodies, prior preeclampsia, prior nephritis, and anti-hypertensive use.

Effect of Educational Tool of Preeclampsia Knowledge: The analysis of the effect of the educational tool on preeclampsia knowledge will be based on the intention-to-treat principle. A Student's t-test will be used to compare the mean preeclampsia questionnaire scores at all visits between the group exposed to the educational tool versus the standard of care group.

Effect of Educational Tool on ASA Adherence: Based on the intention-to-treat principle, investigator will use a Student's t test to analyze the between-group difference using a logarithmic transformation of ARMS scores at the 2rd trimester visit. A logarithmic transformation is used to allow skewed data to approximate a normal distribution. All statistical tests will be 2-sided, and the level of significance will be set at .05.

Sample Size and Power Calculation: The investigator estimates that 40 participants in each group provide at least 80% power, at a 2-sided alpha of .05, to detect a 15% difference in the mean preeclampsia questionnaire score assuming a mean score of 50% with an SD of 10% among women who were unexposed to any educational intervention. As the 6 participating Canadian SLICC centres have a collective number of more than 1 500 SLE women currently enrolled into existing research cohorts, the investigator is confident that the required sample size (total number of required study subjects = 80) will be accrued.

ELIGIBILITY:
Inclusion Criteria

1. Pregnant women with a SLE diagnosis based on the SLICC classification criteria;
2. English and/or French speaking;
3. Followed at participating sites;
4. Gestational age up to 16-6/7 weeks* inclusively
5. Between the ages of 18 and 45 years;
6. Only one pregnancy per woman will be included in the project;
7. Single or multiple intrauterine pregnancies are permitted;
8. Must be participating in the LEGACY Biobank. *Our aim is to recruit subjects under or equal to 12 weeks but we will include pregnancies up to 16-6/7 weeks inclusively

Exclusion Criteria

1. Pregnant women who do not meet the SLE diagnosis based on the SLICC classification;
2. Women who do not speak English or French;
3. Women who are not followed at participating sites;
4. Gestational age at 17 weeks and above
5. Under the age of 18 and over the age of 45;
6. More than one pregnancy per woman will not be included in the project;
7. Women with extrauterine pregnancies;
8. Women who are not participating in the LEGACY Biobank;
9. Women who cannot provide informed consent due to severe illness;
10. Women who are cognitively impaired or incapable of understanding the text written on the consent form;
11. Men are not eligible for this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Change in preeclampsia knowledge in Canadian pregnant women with SLE exposed to an educational tool on preeclampsia versus Canadian women with SLE not exposed to an educational tool | Change from up to and including 12 weeks of pregnancy (baseline) and between 20-24 weeks of pregnancy (second trimester)
  Responses to preeclampsia knowledge questionnaire will be compared at baseline (before randomization) and at second trimester. Questionnaire includes 20 questions, both closed and open ended, regarding preeclampsia implications, symptoms, role of aspirin for its prevention and actions that should be taken if patient experiences preeclampsia symptoms. The questionnaire total score ranges from 0 to 20, with higher score indicating better preeclampsia knowledge. The questionnaire will be scored by 2 independent investigators calculating the number of correct responses.
  Subjects will be randomized in a 1:1 ratio to either patient educational tool or standard of care. SLE specific educational tool consists of sheet displaying the previously developed patient education form on recto. On verso SLE-specific information related to the risk of preeclampsia in SLE pregnancies and the estimated efficacy of ASA in reducing preeclampsia risk in women at high risk are displayed.

SECONDARY OUTCOMES:
Prevalence of ASA use in Canadian pregnant women with SLE receiving standard of care throughout pregnancy | Up to and including 12 weeks of pregnancy, at 20 to 24 weeks of pregnancy, at 30 to 34 weeks of pregnancy, and 8 to 12 weeks after delivery
  At each 4 pregnancy time points, up to and including 12 weeks gestation (baseline), between 20 - 24 weeks (2nd trimester), between 30-34 weeks (3rd trimester) and at 8 to 12 weeks after delivery, patient self-reported ASA use (i.e. current user versus non-user) will be recorded for all participants.
ASA adherence in Canadian pregnant women with SLE in experimental and no intervention groups | Change from up and including 12 weeks of pregnancy (baseline) and between 20-24 weeks of pregnancy (second trimester)
  In participants, the Adherence to Refills and Medications Scale (ARMS) will measure changes in aspirin adherence at baseline and second trimester visit. The ARMS is a validated self-reported questionnaire developed for patients with chronic diseases with low literacy. It includes 12 short and simple questions, each scored 1 ("always") to 4 ("never"), and the total ranges from 12 to 48, with lower scores indicating higher levels of reported adherence. Investigator will define adherence as a continuous variable using the ARMS score and compare the between-group difference using a logarithmic transformation of ARMS scores at the baseline and 2rd trimester visits.
Assessing ASA adherence using a visual analogue scale in Canadian pregnant women with SLE in experimental and no intervention groups | Change from up to and including 12 weeks of pregnancy (baseline) and between 20-24 weeks of pregnancy (second trimester)
  Changes in the visual analogue scale measuring ASA adherence from baseline to second trimester visit.
  On a scale of 0 to 10 where 0 is never and 10 is always, patient-reported adherence to aspirin use will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Vinet, MD/PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Information will be kept between investigators.

REFERENCES:
- [Background] You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. Am J Obstet Gynecol. 2012 May;206(5):431.e1-5. doi: 10.1016/j.ajog.2012.03.006. Epub 2012 Mar 13. PMID 22542120
- [Background] You WB, Wolf M, Bailey SC, Pandit AU, Waite KR, Sobel RM, Grobman W. Factors associated with patient understanding of preeclampsia. Hypertens Pregnancy. 2012;31(3):341-9. doi: 10.3109/10641955.2010.507851. Epub 2010 Sep 22. PMID 20860492
- [Background] Buyon JP, Kalunian KC, Ramsey-Goldman R, Petri MA, Lockshin MD, Ruiz-Irastorza G, Khamashta M. Assessing disease activity in SLE patients during pregnancy. Lupus. 1999;8(8):677-84. doi: 10.1191/096120399680411272. No abstract available. PMID 10568906
- [Background] Bland JM, Altman DG. The use of transformation when comparing two means. BMJ. 1996 May 4;312(7039):1153. doi: 10.1136/bmj.312.7039.1153. No abstract available. PMID 8620137
- [Result] Kripalani S, Risser J, Gatti ME, Jacobson TA. Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value Health. 2009 Jan-Feb;12(1):118-23. doi: 10.1111/j.1524-4733.2008.00400.x. PMID 19911444
- [Derived] Lee JE, Mendel A, Malhame I, Barber MRW, Clarke AE, Fortin PR, Hanly JG, Legge A, Peschken C, Laskin CA, Touma Z, Urowitz MB, Bernatsky S, Vinet E. An educational tool to improve PREeclamPsia knowledge and Aspirin adheRence in lupus prEgnancies: the PREPARE trial. Rheumatology (Oxford). 2025 Nov 1;64(11):5707-5715. doi: 10.1093/rheumatology/keaf334. PMID 40578323